CLINICAL TRIAL: NCT03350880
Title: Effects of Stretching Isquiotibials in Water and on Land in Healthy Adutls for Flexibility: a Randomized Controlled Trial.
Brief Title: Stretching Isquiotibials in Water and on Land in Healthy Adutls
Acronym: Flexibility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do vale do São Francisco (Other)
Responsible Party: Principal Investigator, Rodrigo Gustavo da Silva Carvalho, Master, Universidade Federal do vale do São Francisco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 022017
Record Dates: First submitted 2017-11-18; First posted 2017-11-22 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Muscle Relaxation
Keywords: Passive; Stretching; Water; Proprioceptive Neuromuscular Facilitation (PNF)

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PNF in Water - PNFW (Experimental): Flexibility training was carried out over a period of six weeks, with two sessions per week, totaling 12 sessions.
  Interventions: Other: Flexibility training
- PNF on Land - PNFL (Active Comparator): Flexibility training was carried out over a period of six weeks, with two sessions per week, totaling 12 sessions.
  Interventions: Other: Flexibility training

INTERVENTIONS:
Other: Flexibility training — Flexibility training was carried out over a period of six weeks, with two sessions per week, totaling 12 sessions.
  Other Names: streching training

SUMMARY:
Comparison of therapeutic intervention to gain range of motion at the hip joint within therapeutic in water and on land. Stretching is a therapeutic maneuver used to increase the length of shortened soft tissue structures and thereby gain range of motion; for that, innumerable procedures within Physiotherapy use it for the benefit of patients. The work in question is justified by the need to seek the means that can promote a better performance in the application of the stretching procedure, called Proprioceptive Neuromuscular Facilitation, in a universe of pre-selected volunteers. It is a relevant and feasible study, hoping that its results may benefit future patients, with better results and faster responses. What is the medium that leads to better results in a program using the proprioceptive neuromuscular facilitation technique? Hypotheses: a - Probably the heated aquatic environment, in a range of 32 ° to 36 ° C, will promote a better result, since the heat increases the collagen's distensibility. b - Perhaps the heat, by increasing the excitability threshold of nerve fibers, triggers the "protective reflex" later, which may promote a more vigorous elongation without the protective response. c - Possibly the relaxation promoted in the aquatic environment, could influence the gains obtained in the swimming pool.

DETAILED DESCRIPTION:
Comparison of therapeutic intervention to gain range of motion at the hip joint within therapeutic in water and on land.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 60 years;
* sedentary and who did not perform physiotherapy and physical activity in the last three months;
* clinical and cognitive conditions for swimming pool activities and aerobic exercise; who have not undergone highly complex surgical procedures in the last six months;
* to be able of walking without help equipment and without musculoskeletal or skeletal diseases;
* without contraindications to the practice of exercises; such as: urinary and / or fecal incontinence and dermatological diseases;
* below obesity II with BMI <40.

Exclusion Criteria:

* if they have up to three consecutive fouls during the hydrogymnastics period;
* if they present any adverse effects, such as: allergy or any dermatitis;
* unable to continue the study due to change of address or hospitalization.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-08-28 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
range of motion | six weeks
  range of motion by goniometer

SECONDARY OUTCOMES:
sit and reach test | six weeks
  sit and reach test by wells bank

CONTACTS AND LOCATIONS:
Locations (1):
- Physical Education College, Petrolina, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Papers and abstract congress
Supporting Information: CSR
Time Frame: one year
Access Criteria: age between 18 and 60 years; sedentary and who did not perform physiotherapy and physical activity in the last three months; clinical and cognitive conditions for swimming pool activities and aerobic exercise; who have not undergone highly complex surgical procedures in the last six months; to be able of walking without help equipment and without musculoskeletal or skeletal diseases; without contraindications to the practice of exercises; such as: urinary and / or fecal incontinence and dermatological diseases; below obesity II with BMI <40.

REFERENCES:
- [Result] Ribeiro, Hálisson Alves, et al.
- See also: Effect of proprioceptive neuromuscular facilitation in land and aquatic environments on adult flexibility — https://periodicos.unicesumar.edu.br/index.php/saudpesq/article/view/9938
- Available data/document: Clinical Study Report — https://periodicos.unicesumar.edu.br/index.php/saudpesq/article/view/9938